CLINICAL TRIAL: NCT05197842
Title: A Multicenter, Randomized, Open-lable, Parallel-controlled, Phase I/II Trial to Study Efficacy and Safety of Substitution of Glucocorticoid for BDB-001 Injection in Patients With ANCA-associated Vasculitis
Brief Title: Efficacy and Safety of Substitution of Glucocorticoid for BDB-001 Injection in Patients With Anti-neutrophil Cytoplasmic Antibody(ANCA)-Associated Vasculitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STS-BDB001-07
Record Dates: First submitted 2021-12-02; First posted 2022-01-20 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: ANCA-associated Vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — BDB001; Cyclophosphamide; Glucocorticoids; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group A (Experimental): BDB-001 injection low dose plus reduced dose glucocorticoids in combination with cyclophosphamide
  Interventions: Drug: BDB-001 injection; Drug: Cyclophosphamide; Drug: Glucocorticoids
- Group B (Experimental): BDB-001 injection high dose plus reduced dose glucocorticoids in combination with cyclophosphamide
  Interventions: Drug: BDB-001 injection; Drug: Cyclophosphamide; Drug: Glucocorticoids
- Group C (Active Comparator): Standard dose glucocorticoids in combination with cyclophosphamide
  Interventions: Drug: Cyclophosphamide; Drug: Glucocorticoids
- Group D (Experimental): BDB-001 injection low dose in combination with cyclophosphamide
  Interventions: Drug: BDB-001 injection; Drug: Cyclophosphamide
- Group E (Experimental): BDB-001 injection high dose in combination with cyclophosphamide
  Interventions: Drug: BDB-001 injection; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: BDB-001 injection — Intravenously administered
  Arms: Group A; Group B; Group D; Group E
Drug: Cyclophosphamide — Intravenously administered
Drug: Glucocorticoids — Orally administered
  Other Names: Prednisone
  Arms: Group A; Group B; Group C

SUMMARY:
The aim of the trial is to study the efficacy and safety of treatment with BDB-001 Injection substitution of glucocorticoid in patients with ANCA-associated vasculitis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old≤Age≤75 years old, male or female;
* Diagnosis of granulomatosis with polyangiitis(GPA) or microscopic polyangiitis(MPA)；
* Newly diagnosed or relapsed GPA or MPA that requires treatment with cyclophosphamide(CYC) and glucocorticoids(GCs)；
* Positive test for anti-proteinase 3(PR3) or anti-myeloperoxidase (MPO)；
* Estimated glomerular filtration rate ≥15 mL/minute/1.73 m^2；
* At least 1 major item, or at least 3 non-major items, or at least the 2 renal items on BVAS；

Exclusion Criteria:

* Active tuberculosis infection;
* Severe disease as determined by rapidly progressive glomerulonephritis, alveolar hemorrhage requiring pulmonary ventilation support, rapid-onset mononeuritis multiplex or central nervous system involvement；
* Any other known multi-system autoimmune disease including eosinophilic granulomatosis with polyangiitis (Churg-Strauss), systemic lupus erythematosus, IgA vasculitis (Henoch-Schönlein), rheumatoid vasculitis,anti-glomerular basement membrane disease, or cryoglobulinemic vasculitis；
* HBsAg positive,or HBcAb positive and HBV-DNA positive；
* Received CYC within 3 months before the first administration or Received rituximab(RTX) within 12 months before the first administration；
* Received glucocorticoid shock therapy within 4 weeks before the first administration；
* Received an oral daily dose of a GC of > 10 mg prednisone-equivalent for more than 6 weeks continuously before the first administration；
* Received a anti-tumor necrosis factor and other biological agents treatment within 12 weeks before the first administration；
* Received Continuous dialysis treatment for 12 weeks or more before the first administration; Received Dialysis within 1 week before the first administration;
* Received intravenous immunoglobulin (Ig) or plasma exchange within 4 weeks before the first administration;
* Pregnant or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
The proportion of patients achieving disease complete remission or partial remission assessed by Birmingham Vasculitis Activity Score (BVAS) | 12 weeks

SECONDARY OUTCOMES:
The proportion of patients achieving disease complete remission assessed by Birmingham Vasculitis Activity Score (BVAS) | 12 weeks
Change from baseline in the Birmingham Vasculitis Activity Score (BVAS) | 4 weeks、8 weeks、12 weeks
Change from baseline in the Vasculitis Damage Index (VDI) | 12 weeks
Change from baseline in Estimated glomerular filtration rate (eGFR)、Urinary albumin:creatinine ratio (UACR)、Urine erythrocyte | 4 weeks、8 weeks、12 weeks
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | 0-24weeks
  Safety and tolerability indexes of BDB-001 injection for multiple administration of ANCA-associated vasculitis(AAV) patients
Number of Participants developing anti-BDB-001 antibodies. | 0-24weeks
  Safety and tolerability indexes of BDB-001 injection for multiple administration of ANCA-associated vasculitis(AAV) patients
Area under the plasma concentration versus time curve (AUC) of BDB-001. | 0-12 weeks
  Pharmacokinetic characteristics of BDB-001 injection in AAV patients were characterized based on population pharmacokinetic (PopPK) analysis.
Peak Plasma Concentration (Cmax) of BDB-001 and time to reach Cmax. | 0-12 weeks
  Pharmacokinetic characteristics of BDB-001 injection in AAV patients were characterized based on population pharmacokinetic (PopPK) analysis.
Minimal Plasma Concentration (Cmin) of BDB-001. | 0-12 weeks
  Pharmacokinetic characteristics of BDB-001 injection in AAV patients were characterized based on population pharmacokinetic (PopPK) analysis.
Terminal phase half-life. | 0-12 weeks
  Pharmacokinetic characteristics of BDB-001 injection in AAV patients were characterized based on population pharmacokinetic (PopPK) analysis.
Change from baseline in C5a (mg/dL) concentration. | 0-12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Minghui Zhao, Postdoc, Principal Investigator — Peking University First Hospital
Locations (22):
- China (22):
  - The Second hospital Of Anhui Medical University, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Guangxi Academy of Medical Sciences,The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi Zhuang Autonomous Region (gzar)
  - The Second hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital,Tongji Medical college of Hust, Wuhan, Hubei
  - Xiangya Hospital Central South University (Nephrology Department), Changsha, Hunan
  - Xiangya Hospital Central South University(Rheumatism Immunity Branch), Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shengyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia Hui Autonomous Region(NHAR)
  - Zhongshan hospital,Fudan University, Shanghai, Shanghai Municipality
  - Xijing Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No